CLINICAL TRIAL: NCT03150264
Title: The Comparison of Pressure-controlled Ventilation and Pressure-controlled Ventilation Volume-guaranteed on Respiratory Dynamics and Clinical Outcome in Patients Undergoing Bariatric Surgery: Prospective Clinical Study
Brief Title: Prospective Clinical Study of PCV and PCV-VG in Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wu Pan, Principal Investigator, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: clinical review (2016) (397)
Record Dates: First submitted 2017-04-21; First posted 2017-05-12 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Bariatric Surgery; Mechanical Ventilation
Keywords: lung protective ventilation strategies; obesity
MeSH Terms: conditions — Obesity | interventions — Hematocrit

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCV-VG+PEEP5cmH₂O (Experimental): Patients in this group are ventilated with pressure-controlled ventilation volume-guaranteed mode. And we use PEEP of 5cmH₂O to open the collapsed alveoli.
  Interventions: Device: PCV-VG, PEEP5cmH₂O
- PCV+PEEP5cmH₂O (Active Comparator): Patients in this group are ventilated with pressure-controlled ventilation mode. And we use PEEP of 5cmH₂O to open the collapsed alveoli.
  Interventions: Device: PCV, PEEP5cmH₂O

INTERVENTIONS:
Device: PCV-VG, PEEP5cmH₂O — This is an innovative ventilation mode developed in recent years. The preset tidal volume help the machine modify inspiratory pressures and compensate the decrease of lung compliance.
  Arms: PCV-VG+PEEP5cmH₂O
Device: PCV, PEEP5cmH₂O — This is a traditional ventilation mode used in obese patients in the past.
  Arms: PCV+PEEP5cmH₂O

SUMMARY:
This study compares the two mechanical ventilation strategies in obese patients undergoing bariatric surgery: pressure-controlled ventilation(PCV) and pressure-controlled ventilation volume-guaranteed（PCV-VG). This is a randomized controlled trial with a sample size of 100 patients whose body mass index(BMI) is over 30kg/m².

DETAILED DESCRIPTION:
With the development of economy and changing of life style, obesity is becoming a common phenomenon. More and more obese patients are undergoing bariatric surgery every year.

Obesity results in a series of physiological changes particularly the respiratory system. The decrease of lung compliance and the limited total lung capacity, vital capacity, functional residual capacity are all contributed to intraoperative hypoxemia and postoperative lung complications. Presently study mainly discuss lung protective ventilation strategies from four aspects: tidal volume,ventilation modes,positive end-expiratory pressures and lung recruitment maneuvers.

This prospective study will compare two ventilation modes in obese patients undergoing bariatric surgery:pressure-controlled ventilation(PCV) and pressure-controlled ventilation volume-guaranteed（PCV-VG).

The total of 100 patients will be divided into two groups randomly. The patients will be ventilated with PCV or PCV-VG modes plus positive end expiratory pressure (PEEP) of 5cmH2O throughout the whole operation.

The respiratory and hemodynamic parameters in six time points will be recorded, and the postoperative chest computerized tomography (CT) will be checked to identify the postoperative lung complications.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥30kg/m²
* ASA classification II-III
* Bariatric surgery

Exclusion Criteria:

* Patients combined restrictive or obstructive lung diseases,pneumonia, bullae of lung ; patients after pneumonectomy
* Patients combined with other severe internal medicine diseases
* duration of pregnancy or suckling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic lung compliance measure | three hours
  Dynamic lung compliance can be calculated based on tidal volume,peak inspiratory pressure and PEEP. 10minutes after induction,10minutes after pneumoperitoneum,60minutes after pneumoperitoneum and 10minutes after pneumoperitoneum release will be recorded.

SECONDARY OUTCOMES:
Postoperative lung complications | five days
  Lung complications mainly contains pneumonia,atelectasis,pleural fluid. The investigator compare the preoperative chest CT with the postoperative chest CT and follow-up participants until participants leave hospital.
the risk factors of postoperative lung complications | five days
  risk factors may include age, gender, BMI, ventilation duration, etc

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Liang, doctor, Study Director — Huashan Hospital
Locations (1):
- Fudan University Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD is available only when we finish or publish the study. Please contact me via e-mail of this account.
Supporting Information: Study Protocol, CSR
Time Frame: The information is available only when we finish or publish the study. Please contact me via e-mail of this account.
Access Criteria: Open for the clinical researchers

REFERENCES:
- [Result] Dion JM, McKee C, Tobias JD, Sohner P, Herz D, Teich S, Rice J, Barry ND, Michalsky M. Ventilation during laparoscopic-assisted bariatric surgery: volume-controlled, pressure-controlled or volume-guaranteed pressure-regulated modes. Int J Clin Exp Med. 2014 Aug 15;7(8):2242-7. eCollection 2014. PMID 25232415
- [Result] Aldenkortt M, Lysakowski C, Elia N, Brochard L, Tramer MR. Ventilation strategies in obese patients undergoing surgery: a quantitative systematic review and meta-analysis. Br J Anaesth. 2012 Oct;109(4):493-502. doi: 10.1093/bja/aes338. PMID 22976857
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4161575/